CLINICAL TRIAL: NCT04229381
Title: Resiliency Among Older Adults Receiving Lung Cancer Treatment (ROAR-LCT): Physical Therapy and Progressive Muscle Relaxation in Improving Physical Performance and Mood in Older Patients With Stage IIIA-B or IV Lung Cancer Undergoing Treatment
Brief Title: Resiliency Among Older Adults Receiving Lung Cancer Treatment
Acronym: ROAR-LCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Carolyn Presley, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-19115; NCI-2019-04722 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R03AG064374 (NIH)
Record Dates: First submitted 2019-11-26; First posted 2020-01-18 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-10

CONDITIONS: Advanced Lung Carcinoma; Extensive Stage Lung Small Cell Carcinoma; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8; Unresectable Lung Carcinoma; Unresectable Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Physical Therapy Modalities; Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (physical therapy, muscle relaxation) (Experimental): Patients participate physical therapy sessions consisting of cardiovascular and resistance training exercises in person or online and also undergo progressive muscle relaxation sessions once weekly for up to 12 weeks.
  Interventions: Procedure: Physical Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Relaxation Therapy

INTERVENTIONS:
Procedure: Physical Therapy — Undergo physical therapy
  Other Names: Physiatric Procedure; Physical Medicine Procedure; Physical Therapeutics; Physical Therapy Procedure; Physiotherapy; Physiotherapy Procedure; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Relaxation Therapy — Undergo progressive muscle relaxation

SUMMARY:
This trial studies how well physical therapy and progressive muscle relaxation works in improving physical performance and mood in older patients with stage IIIA-B or IV lung cancer who are undergoing treatment. Improving physical performance and mood may help older patients maintain an independent lifestyle by helping to improve their resilience, the ability to bounce back to normal functioning after a stressor or intervening health event such as treatment or disease progression. Giving physical therapy and progressive muscle relaxation may work in improving symptoms and quality of life in patients with lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of a novel, weekly supervised virtual health-assisted physical therapy plus relaxation intervention delivered to older adults with advanced thoracic malignancy (N=20).

OUTLINE:

Patients participate physical therapy sessions consisting of cardiovascular and resistance training exercises in person or online and also undergo progressive muscle relaxation sessions once weekly for up to 12 weeks.

After completion of study therapy, patients are followed up at 24 weeks, and then periodically for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with advanced lung cancer: unresectable stage IIIA, IIIB, or stage IV non-small cell lung cancer (NSCLC) or extensive stage small cell lung cancer (SCLC).
* Intent to receive treatment from the Ohio State University Comprehensive Cancer Center (OSUCCC) Thoracic Oncology Clinic.
* Willingness to participate and adhere to the study intervention program.
* Ability to understand and willingness to sign an informed consent document (or indicate approval or disapproval by another means).

Exclusion Criteria:

* Prisoners are excluded from participation.
* There is NO exclusion criteria pertaining to Eastern Cooperative Oncology Group (ECOG) performance status, laboratory values, prior cancer diagnoses, presence of comorbidities or brain metastases.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn J Presley, MD, MHS, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive Care (Physical Therapy, Muscle Relaxation)
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (Physical Therapy, Muscle Relaxation)
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 71.9 [60 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
Lung Cancer Type [Count of Participants; unit: Participants]
  Non-Small Cell Lung Cancer (NSCLC) | 15
  Small Cell Lung Cancer (SCLC) | 3

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rates
Description: Recruitment rates will be defined as the proportion of screened older adults accrued relative to those approached in the Ohio State University Comprehensive Cancer Center (OSUCCC) Thoracic Oncology Clinic. Successful recruitment rates will be defined as >= 50% of older adults (>= 60 years) approached agree to participate.
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Physical Therapy, Muscle Relaxation)
Number analyzed (Participants) | 18
Participants | 11

2. Primary Outcome: Adherence Rate
Description: Study adherence will be defined as the completion of >= 70% of the program sessions, repeated assessments, and collection of bio specimens either at the end of the study period or death, whichever occurs first.
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Physical Therapy, Muscle Relaxation)
Number analyzed (Participants) | 18
Participants | 11

3. Primary Outcome: Retention Rates
Description: Retention rates will be defined as the percentage of participants not lost to follow-up.
Time Frame: Up to 24 weeks
Population: 22 patients were consented and enrolled. 4 of the patients that underwent informed consent withdrew from the study prior to completing any study activities. This leaves a total of 18 evaluable participants analyzed for study adherence and retention. Acceptability was defined as completing at least 70 percent of all study visits and not lost to follow up. 2 patients withdrew from the study after beginning the ROAR intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Physical Therapy, Muscle Relaxation)
Number analyzed (Participants) | 18
Participants | 16

4. Secondary Outcome: Functional Trajectories
Description: Evaluated using generalized linear mixed models (GLMMS). GLMMs can determine whether factors affect all patient trajectories in similar ways or whether they affect individual trajectories differently. To allow for possible changes in functional status over time (e.g., a change-point analysis) the 'segmented' package in R will be used. Participants' functional status scores will be modeled using a segmented mixed model with random change points. Estimating the change point identifies the point in time that patients' functional status scores change during the 12-months post-diagnosis.
Time Frame: At 12 months
Population: Data not collected and analyzed
Arm/Group | Supportive Care (Physical Therapy, Muscle Relaxation)
Number analyzed (Participants) | 0

5. Secondary Outcome: Factors Associated With Resiliency
Description: Evaluated using GLMMS. Resiliency will be defined as the ability to maintain or regain at least 50% of baseline functional status at any point during the 12 months after diagnosis with specific emphasis at 3 and 6-months post- the start of treatment. The association between resiliency and clinical factors will be evaluated with appropriate statistical techniques for the specific measure (e.g. Chi-square tests will compare categorical variables between participants demonstrating resiliency vs. worsening functional status; a two-sample t-test or Wilcoxon Rank Sum test will compare continuous variables).
Time Frame: Up to 12 months
Population: Data not collected and analyzed
Arm/Group | Supportive Care (Physical Therapy, Muscle Relaxation)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: A minimum of 12 weeks or through study completion, an average of 1 year
Description: Adverse event information was collected for study patients form baseline through study completion utilizing the CTCAE Version 4.0 to determine the severity of the event through study completion.
Arm/Group | Supportive Care (Physical Therapy, Muscle Relaxation)
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
Study opened in February of 2020 and COVID-19 lockdown in Ohio occurred in March of 2020. We had participants already in this first month of accrual who did decide to dropout due to COVID-19 related concerns. The study design was modified as most patients were being seen via virtual health for standard oncology care visits. The first and final intervention sessions were in-person with the remainder conducted via virtual health.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT04229381/Prot_SAP_001.pdf
  • Informed Consent Form (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT04229381/ICF_002.pdf